CLINICAL TRIAL: NCT04944173
Title: A Phase II Study of Circulating Tumor DNA Directed Consolidation Durvalumab (MEDI4736) Following Induction and Concurrent Durvalumab with SABR for Stage I NSCLC. SCION: SABR and Checkpoint Inhibition of NSCLC
Brief Title: SCION: SABR and Checkpoint Inhibition of NSCLC
Acronym: SCION
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Overestimated pool of eligible patients and the potential participants either declined participation or did not meet eligibility criteria.
Sponsor: University of British Columbia (Other)
Collaborators: AstraZeneca (Industry); Ozmosis Research Inc. (Industry)
Responsible Party: Principal Investigator, Islam Mohamed, Clinical Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H21-00994; OZM-119 (Other: Ozmosis Research (CRO))
Record Dates: First submitted 2021-06-17; First posted 2021-06-29 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Non Small Cell Lung Cancer; Carcinoma, Non-Small-Cell Lung; Non-small Cell Lung Cancer Stage I; Lung Cancer; Lung Cancer Stage I; Lung Adenocarcinoma, Stage I; Lung Squamous Cell Carcinoma Stage I
Keywords: durvalumab; Imfinzi; MEDI4736; MEDI-4736; Circulating Tumor DNA; Cell-Free Tumor DNA; Minimal Residual Disease; Stereotactic Radiation Therapy; Stereotactic Body Radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Adenocarcinoma of Lung; Neoplasm, Residual | interventions — durvalumab; Radiosurgery

STUDY DESIGN:
Intervention Model Description: Study subjects will be analyzed as a single cohort with respect to the primary outcome, with comparison to historical controls. Treatment assignment based on biomarker status after initial treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- MRD Negative (Experimental): All subjects will receive four cycles of durvalumab with SABR concurrent at cycle 2, then will be evaluated for MRD. Subjects in this arm have no detectable ctDNA at MRD landmark and will receive no further therapy.
  Interventions: Drug: Durvalumab; Radiation: Stereotactic Body Radiotherapy; Diagnostic Test: Circulating Tumor DNA assay
- MRD Positive, no further therapy (Experimental): All subjects will receive four cycles of durvalumab with SABR concurrent at cycle 2, then will be evaluated for MRD. Subjects in this arm have detectable ctDNA at MRD landmark and are randomized to no further therapy.
  Interventions: Drug: Durvalumab; Radiation: Stereotactic Body Radiotherapy; Diagnostic Test: Circulating Tumor DNA assay
- MRD Positive, consolidation durvalumab (Experimental): All subjects will receive four cycles of durvalumab with SABR concurrent at cycle 2, then will be evaluated for MRD. Subjects in this arm have detectable ctDNA at MRD landmark and are randomized to eight additional cycles of durvalumab
  Interventions: Drug: Durvalumab; Radiation: Stereotactic Body Radiotherapy; Diagnostic Test: Circulating Tumor DNA assay

INTERVENTIONS:
Drug: Durvalumab — Subjects will receive durvalumab 1500mg IV every four weeks for four cycles, undergo assessment for residual disease, then a subset of subjects will receive an additional eight cycles of durvalumab.
  Other Names: MEDI4736; Imfinzi
Radiation: Stereotactic Body Radiotherapy — Subjects will receive stereotactic radiation therapy concurrent with cycle 2 of durvalumab to a dose of 48Gy in four fractions. Fractionation may be modified for central tumors.
  Other Names: Stereotactic Radiation; Stereotactic Radiation Therapy
Diagnostic Test: Circulating Tumor DNA assay — After four cycles of durvalumab, subjects will be evaluated at the MRD Landmark for residual ctDNA to determine subsequent treatment assignment.
  Other Names: AVENIO ctDNA surveillance assay; MRD Landmark assay

SUMMARY:
The SCION Trial is a clinical trial in patients with early stage non-small cell lung cancer. The purpose of the trial is to investigate whether it is safe and effective to combine standard radiation treatment with a drug called durvalumab, a type of immunotherapy. In addition, the study will use a blood test to look for cancer cell DNA to determine how long treatment with durvalumab should last. Both the use of durvalumab and the use of the blood test are new strategies for managing early stage non-small cell lung cancer.

DETAILED DESCRIPTION:
PURPOSE The intent of the study is to determine whether disease control in early non-small cell lung cancer (NSCLC) achieved by stereotactic ablative body radiotherapy (SABR) can be augmented locally, regionally, and distantly by safely combining it with durvalumab. Moreover, the study will assess whether patients who are likeliest to benefit from extended treatment with durvalumab can be predicted by assaying for molecular residual disease (MRD) after initial treatment using the AVENIO assay for circulating tumor DNA (ctDNA).

HYPOTHESIS Combining SABR and Durvalumab in patients with T1-2 N0 M0 NSCLC reduces the overall relapse rate at 18 months by 50% compared with historical controls treated with SABR alone, from 19.3% to 9.7%.

OBJECTIVES Primary

• To determine the overall relapse rate at 18 months in patients with T1-2 N0 M0 NSCLC treated with SABR and Durvalumab.

Secondary

* To determine rates of Local Relapse, Regional Nodal Relapse, Distant Relapse, and Second Primary Lung Cancer in patients with T1-2 N0 M0 NSCLC treated with SABR and Durvalumab.
* To determine rates of Overall Survival, Cause-Specific Survival, and Relapse Free Survival in patients with T1-2 N0 M0 NSCLC treated with SABR and Durvalumab
* To determine rates of pneumonitis, immune-related toxicity, adverse events, serious adverse events in patients with T1-2 N0 M0 NSCLC treated with SABR and Durvalumab.
* To determine the rate of MRD detection using the AVENIO ctDNA assay in patients with T1-2 N0 M0 NSCLC treated with SABR and Durvalumab.
* To compare clinical outcomes between patients with detectable versus undetectable MRD using the AVENIO ctDNA assay following treatment with SABR and Durvalumab.
* To compare clinical outcomes between patients with detectable MRD using the AVENIO ctDNA assay following treatment with SABR and Durvalumab who receive extended Durvalumab versus no further therapy.

STUDY DESIGN Subjects who meet the eligibility criteria will be candidates for enrolment. All subjects will receive one infusion of Durvalumab every 4 weeks for four cycles (4 weeks = 1 cycle), with SABR delivered concurrently with cycle 2. Subjects will be assessed at baseline using the AVENIO assay initially on tumor tissue. This will allow the subsequent evaluation for molecular residual disease (MRD) following cycle 4 to be tumor-informed, and ultrasensitive. Subjects with no detectable ctDNA at the MRD assessment will receive no further therapy. Subjects with detectable ctDNA at the MRD assessment will be randomized to receive either no further therapy or 8 additional cycles of q4w Durvalumab. Safety will be evaluated by recording the occurrence of adverse events, serious adverse events, and laboratory abnormalities, with special attention to pneumonitis and immune-related toxicity.

Future research will be enabled through the collection of biospecimens. Subjects will separately consent to the optional collection of these biospecimens. Blood samples collected for this purpose at multiple timepoints (0, 4, 12, 24 months) will be archived in a biorepository created for this study operated by the BC Cancer Tumour Tissue Repository (Victoria, BC). Stool samples collected for this purpose at multiple timepoints (0, 4, and 12 months) will be archived in the Oncomicrobiome Repository (Montreal, QC).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be competent, >18yo at time of study entry, and capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization (e.g., Health Insurance Portability and Accountability Act in the US, European Union [EU] Data Privacy Directive in the EU) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
2. Patients with histological diagnosis of NSCLC, all histological sub-types are eligible
3. Body weight >30kg
4. ECOG Performance status (PS) 0-2.
5. Tumor stage T1-2 (≤5cm) N0 M0 (8th Edition of the TNM Classification for Lung Cancer) based on CT chest/abdomen, FDG-PET within 12 weeks of enrolment, and, where performed, EBUS-guided biopsy of hilar or mediastinal nodes within 8 weeks of enrolment.
6. Subject deemed medically inoperable, or subject deemed operable but declines surgery following surgical assessment.
7. Peripheral (outside a 2cm radius proximal bronchial tree) and central (within 2cm, but neither abuts nor invades proximal bronchial tree) tumors permitted.
8. Screening laboratory values for organ function must meet the following criteria within 14 days prior to cycle 1 day 1:

   * Bone Marrow: Absolute neutrophils ≥ 1.5 x 10^9/L; Platelets ≥ 100 x 10^9/L; Hemoglobin ≥ 90 g/L
   * Kidney: Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

   Males:

   Creatinine CL (mL/min) = Weight (kg) x (140 - Age)

   ÷ 72 x serum creatinine (mg/dL)

   Females:

   Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85

   ÷ 72 x serum creatinine (mg/dL)
   * Liver: AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal
   * serum bilirubin ≤ 1.5 X ULN
   * Cardiac: LVEF ≥ 50%
9. No prior chemotherapy or planned adjuvant chemotherapy is allowed
10. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

    * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
    * Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
11. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
12. Must have a life expectancy of at least 12 weeks.

Exclusion Criteria:

1. Any patient with malignancy which cannot be reliably defined on the treatment planning CT scan due to adjacent opacification from effusion, consolidation, or atelectasis.
2. History of allogenic organ transplantation.
3. History of active primary immunodeficiency
4. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

   1. Patients with vitiligo or alopecia
   2. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
   3. Any chronic skin condition that does not require systemic therapy
   4. Patients without active disease in the last 5 years may be included but only after consultation with the study physician
   5. Patients with celiac disease controlled by diet alone
5. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
6. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C and HIV. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
7. History of another primary malignancy except for:

   1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence
   2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
   3. Adequately treated carcinoma in situ without evidence of disease
8. Participation in another clinical study with an investigational product during the last 2 months
9. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
10. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

    1. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
    2. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician.
11. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
12. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug
13. Previous radiotherapy to the chest or mediastinum. Subjects who have had previous breast radiotherapy may be eligible at the discretion of the Sponsor.
14. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP.
15. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
16. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart).
17. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

    1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    2. Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent
    3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
18. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy.
19. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
20. Prior randomization or treatment in a previous durvalumab clinical study regardless of treatment arm assignment.
21. Patients who have received prior anti-PD-1, anti PD-L1 or anti CTLA-4:

    1. Must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy.
    2. All AEs while receiving prior immunotherapy must have completely resolved or resolved to baseline prior to screening for this study.
    3. Must not have experienced a ≥Grade 3 immune related AE or an immune-related neurologic or ocular AE of any grade while receiving prior immunotherapy. NOTE: Patients with endocrine AE of ≤Grade 2 are permitted to enroll if they are stably maintained on appropriate replacement therapy and are asymptomatic.
    4. Must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE, not have experienced recurrence of an AE if re-challenged, and not currently require maintenance doses of > 10 mg prednisone or equivalent per day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Overall Risk of Relapse | 18 months
  Fraction of subjects experiencing relapse at 18 months following initial therapy

SECONDARY OUTCOMES:
Radiographic Response by RECIST criteria | 6 months (CT) and 12 months (PET/CT)
  Evaluation of radiographic response by CT and PET/CT
Local Relapse | 18 months
  Recurrence at irradiated primary tumor site
Regional Nodal Relapse | 18 months
  Recurrence in a hilar or mediastinal node
Distant Metastatic Relapse | 18 months
  Recurrence in a distant metastatic site
Overall Survival | 18 months
  Proportion of subjects remaining alive
Cause-Sepcific Survival | 18 months
  Proportion of subjects surviving lung cancer in the absence of other causes of death
Relapse Free Survival | 18 months
  Proportion of subjects surviving without relapse
Second Primary Lung Cancer rate | 18 months
  Proportion of subjects diagnosed with a second primary lung cancer at a site beyond the treatment volume
Molecular Residual Disease rate | 6 months
  Proportion of subjects with detectable ctDNA on MRD Landmark assay
Adverse Events | 18 months
  Number and severity of adverse events
Serious Adverse Events | 18 months
  Number and severity of serious adverse events
Pneumonitis | 12 months
  Number and severity of subjects experiencing pneumonitis
Immune-related Adverse Events | 18 months
  Number and severity of subjects experiencing immune-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Islam Mohamed, MD, Principal Investigator — BC Cancer
Locations (5):
- Canada (5):
  - BC Cancer--Kelowna, Kelowna, British Columbia
  - BC Cancer--Surrey, Surrey, British Columbia
  - BC Cancer--Vancouver, Vancouver, British Columbia
  - BC Cancer--Victoria, Victoria, British Columbia
  - Juravinski Cancer Centre, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.